CLINICAL TRIAL: NCT06854445
Title: Phase II Clinical Trial of TQB2825 Injection Combined With Chemotherapy in Subjects With Relapsed/Refractory Diffuse Large B-cell Lymphoma
Brief Title: Clinical Trial of TQB2825 Injection Combined With Chemotherapy in Subjects With Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chia Tai Tianqing Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2825-II-01
Record Dates: First submitted 2025-02-26; First posted 2025-03-03 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-11

CONDITIONS: Diffuse Large Cell B-lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Gemcitabine; Injections; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2825 Injection + Gemcitabine Hydrochloride for Injection + Oxaliplatin for Injection (Experimental): The subject received TQB2825 injection, gemcitabine hydrochloride for injection, and oxaliplatin for injection.
  Interventions: Drug: TQB2825 Injection + Gemcitabine Hydrochloride for Injection + Oxaliplatin for Injection

INTERVENTIONS:
Drug: TQB2825 Injection + Gemcitabine Hydrochloride for Injection + Oxaliplatin for Injection — Drug: TQB2825 Injection + Gemcitabine Hydrochloride for Injection + Oxaliplatin for Injection;
  Other Name:
  Gemcitabine Hydrochloride for Injection, Zefei; Oxaliplatin for Injection, Aihen
  TQB2825 injection is Cluster of Differentiation 3 (CD3) and and Cluster of Differentiation 20 (CD20) bispecific antibody; Gemcitabine hydrochloride for injection is a cell cycle-specific antimetabolite; Oxaliplatin for Injection is a platinum chemotherapy drug.

SUMMARY:
The purpose of this study is to assess the preliminary efficacy of TQB2825 in combination with chemotherapy in subjects with diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily participate in this study, sign the informed consent form, and have good compliance;
* Age ≥18 years (calculated from the date of informed consent);
* Eastern Cooperative Oncology Group (ECOG) score 0 ~ 2 points;
* Expected survival greater than 12 weeks;
* Histological or cytological diagnosis of diffuse large B-cell lymphoma in accordance with the World Health Organization (WHO) diagnostic criteria in 2022;
* Pathological diagnosis results containing CD20 positive expression and Myc rearrangement negative after anti-CD20 treatment must be provided;
* Subjects with relapsed or refractory diffuse large B-cell lymphoma who have received at least 1 line of systemic therapy;
* Not suitable for hematopoietic stem cell transplantation;
* According to the Lugano criteria in 2014, there is at least one measurable lesion, that is, the long diameter of lymph node lesions > 15 mm or extranodal lesions > 10 mm according to CT cross-sectional images; Positron emission tomography - computerized tomography (PET-CT) scan shows PET positive;
* Laboratory tests meet specific criteria;
* Adopt effective contraceptive measures;

Exclusion Criteria:

* Subjects who had or currently had other malignant tumors within 5 years prior to the first dose;
* Previous or current involvement or suspected involvement of the central nervous system by lymphoma;
* Failure to recover from adverse reactions to Common Terminology Criteria for Adverse Events version 5.0 (CTCAEv5.0) criteria ≤ grade 1 from previous treatment;
* History of previous anti-tumor treatment:

  1. previous use of other antibody drugs targeting CD3 and CD20 at the same time;
  2. received Chimeric Antigen Receptor T-Cell Immunotherapy (CAR-T) therapy, or other immune cell therapy, or autologous hematopoietic stem cell transplantation (auto-HSCT) within 3 months before the first dose;
  3. previous treatment with R-GemOx or GemOx;
  4. received chemotherapy, immunotherapy, monoclonal antibody therapy 4 times before the first dose, 2 times received radiotherapy or small molecule targeted drugs, or subjects who are still within 5 half-lives of the drug, the washout period is calculated from the end time of treatment;
  5. received treatment with Chinese patent medicines with clear anti-tumor indications in the package insert of National Medical Products Administration (NMPA)-approved drugs 2 times before the first dose;
* Subjects who have undergone major surgical treatment, significant traumatic injury, or expected major surgery during the study treatment period within 4 weeks prior to the first use of medication, or have long-term untreated wounds or fractures;
* Subjects who experience any bleeding or bleeding events ≥ Common Terminology Criteria Adverse Event (CTC AE) grade 3 within 4 weeks prior to the first administration;
* Hyperactive/venous thrombotic events within 6 months prior to first dose,Such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism or any other history of severe thromboembolism;
* Clinically significant uncontrolled pleural effusion, ascites and more than moderate pericardial effusion requiring repeated drainage;
* Decompensated cirrhosis (Child-Pugh class B or C liver function) and active hepatitis;
* Pulmonary disease, including any of the following: 1) with or without current pneumonitis requiring corticosteroid therapy; 2) with or suspected chronic obstructive pulmonary disease (COPD), and forced expiratory volume in 1 second (FEV1) < 60% (predicted);
* Brain or mental disorders;
* Have major cardiovascular disease;
* Active or uncontrolled infection (≥ CTCAE grade 2 infection), including bacterial, fungal or viral infections including but not limited to active pneumonia, syphilis and tuberculosis.
* Unexplained fever > 38.5℃ during screening or before the first dose;
* Renal failure requiring hemodialysis or peritoneal dialysis, previous history of nephrotic syndrome;
* History of immunodeficiency, including HIV-positive or other acquired, congenital immunodeficiency diseases;
* Have or have had prior autoimmune disease requiring treatment.
* Prepare to undergo or have previously received organ transplantation, or have a significant host transplant response, or have previously received allogeneic hematopoietic stem cell transplantation; 19、Need to receive systemic immunosuppressive therapy;
* Known or suspected history of hemophagocytic syndrome (HLH);
* Known hypersensitivity to excipient components of the study drug.
* Subjects who participated in other anti-tumor clinical trials within 4 or 5 half-lives before the first dose.
* Any condition that, in the judgment of the investigator, would jeopardize the safety of the subject or prevent the subject from completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CR rate) | 1 year
  Percentage of subjects with complete (CR) per 2014 Lugano criteria.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 1 year
  Percentage of subjects with complete (CR) or partial response (PR) according to 2014 Lugano Criteria.
Progression-free survival (PFS) | 1 year
  Time from randomization or first dose to disease progression or death from any cause, whichever occurs first, as determined by the 2014 Lugano Criteria.
Duration of Response (DOR) | 1 year
  The time from first achievement of response, to disease progression or death from any cause, whichever comes first, was determined according to the 2014 Lugano criteria.
Time to Response (TTR) | 1 year
  Time from randomization or first dose of trial drug to the first evaluation of PR or CR, whichever occurs first.
Overall survival (OS) | 3 years
  From randomization to the time of death from any cause.
Half-life (t1/2) | Pre-dose, 5 minutes, 24, 72, 120 and 168 hours post dose on day 1 of cycles 2, 4; pre-dose, 5 minutes post dose on day 1 of cycles 3, 8; once at the end of treatment, each cycle is 21 days
  Time required for the amount of drug in the body or blood concentration to be reduced by half.
Area under the plasma concentration-time curve (AUC0-last) | Pre-dose, 5 minutes, 24, 72, 120 and 168 hours post dose on day 1 of cycles 2, 4; pre-dose, 5 minutes post dose on day 1 of cycles 3, 8; once at the end of treatment, each cycle is 21 days
  Area under the dynamic curve of plasma concentration over time.
Apparent clearance (CL) | Pre-dose, 5 minutes, 24, 72, 120 and 168 hours post dose on day 1 of cycles 2, 4; pre-dose, 5 minutes post dose on day 1 of cycles 3, 8; once at the end of treatment, each cycle is 21 days
  The rate at which the drug is cleared from the body.
Apparent volume of distribution at terminal phase (Vz) | Pre-dose, 5 minutes, 24, 72, 120 and 168 hours post dose on day 1 of cycles 2, 4; pre-dose, 5 minutes post dose on day 1 of cycles 3, 8; once at the end of treatment, each cycle is 21 days
  The volume of body fluid required to distribute the drug in the body according to the plasma drug concentration at this time after the drug distribution in the plasma and tissues has reached equilibrium.
Trough plasma concentration (Cmin) | Pre-dose, 5 minutes, 24, 72, 120 and 168 hours post dose on day 1 of cycles 2, 4; pre-dose, 5 minutes post dose on day 1 of cycles 3, 8; once at the end of treatment, each cycle is 21 days
  Maximum blood concentration achieved by drug administration.
Anti-drug antibody (ADA ) incidence | 2 years
  Immunogenicity test: Anti-drug antibody (ADA ) incidence.

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Affiliated Cancer Hospital and insititute Guangzhou Medical University, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital (HBCH), Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong cancer hospital, Jinan, Shandong
  - Weihai Central Hospital, Weihai, Shandong
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Sichuan Provincal People's Hospital, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - THE First Affiliated Hospital ZheJiang University School of Medicine, Hangzhou, Zhejiang